CLINICAL TRIAL: NCT00225004
Title: Low-energy Fracture of the Wrist (Colles Fracture) and Osteoporosis. A Ten Year Follow-up and a Prospective Study
Brief Title: Osteoporosis and Colles Fracture
Status: Terminated | Type: Observational
Why Stopped: Recruiting problems
Sponsor: Northern Orthopaedic Division, Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: ON-06-002-AJ
Record Dates: First submitted 2005-09-21; First posted 2005-09-23 (Estimated); Last update posted 2014-04-03 (Estimated); Status verified 2014-04

CONDITIONS: Previous or Actual Colles Fracture
Keywords: Colles Fracture; Osteoporosis; BMD; Quality assurance
MeSH Terms: conditions — Colles' Fracture; Osteoporosis | interventions — Absorptiometry, Photon

STUDY DESIGN:
Time Perspective: Retrospective

INTERVENTIONS:
Procedure: DEXA scan — orto

SUMMARY:
The primary purpose of the retrospective study is to determine the incidence of osteoporosis in women with previous Colles Fracture. Secondly, to determine to which extent Colles Fracture has led to a diagnosis and/or treatment of osteoporosis.

The primary purpose of the prospective study is to determine the incidence of osteoporosis in women with an actual Colles Fracture. Secondly, to investigate the consistency between prospective and retrospective data.

DETAILED DESCRIPTION:
Colles Fracture is known to be connected to decreased bone mineral density (BMD). Thus, it can be an early sign of osteoporosis and therefore an increased risk of new fractures.

The results of earlier studies have not been unambiguous in the respect of what extent decreased BMD in the wrist of women with Colles Fracture is synonymous of osteoporosis in the spine and the hip.

An earlier enquiry to the Danish Orthopedic Departments in 1995 showed that only 18 % of the departments diagnosed or referred patients with possible osteoporosis.

The two study designs enhance the possibilities of evaluating the relevance of Low Energy Fractures in the wrist to avoid new fractures and their relation to bone mineral density.

The results could also be a useful tool in quality assurance of the osteoporosis diagnostics.

ELIGIBILITY:
Inclusion Criteria:

Colles Fracture Women over 40 years Informed consent-

Exclusion Criteria:

High Energy Fracture Deceases or conditions that makes the participant unable to contribute to the investigation-

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: years
Sampling Method: Non-Probability Sample
Dates: Start 2004-07

PRIMARY OUTCOMES:
The incidence of Osteoporosis ten years after a Colles Fracture | years
The incidence of Osteoporosis in women with an actual Colles Fracture | years

CONTACTS AND LOCATIONS:
Overall Officials: Klaus K Pedersen, doctor, Principal Investigator — Dept. of Orthopedic Northern Jutland Counties, Denmark; Klaus K Pedersen, doctor, Principal Investigator — Department of Orthopedic surgery, Northern Jutland Counties, Denmark
Locations (2):
- Denmark (2):
  - The department of Orthopedic surgery Northern Jutland Counties, Denmark, Aalborg, Jutland
  - Northern Orthopaedic Division, Klinik Aalborg, Aalborg, Northern Jutland